CLINICAL TRIAL: NCT03085316
Title: Electrical Stimulation of Laryngeal Muscles to Restore Glottal Opening in Patients with Bilateral Vocal Fold Paralysis
Brief Title: Laryngeal Pacing Study
Acronym: BVFP IDE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was halted early as grant funding was awarded for a new study, which was opened in place of this one.
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, David Zealear, PhD, Professor, Department of Otolaryngology, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 141242
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Bilateral Vocal Fold Paralysis (BVFP)
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: All patients who meet eligibility will undergo device implantation surgery and follow up per protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Investigational Device (Experimental): Patient who meets eligibility to be implanted with the St. Jude Medical Infinity™ Implantable Pulse Generator System (P140049), St. Jude Medical Infinity™ Deep Brain Stimulation (DBS) Directional Lead and Extension (P140009), Swift-Lock™ Anchor (K092371), Butterfly anchor (P140009), manufactured by St. Jude Medical, Inc.
  Interventions: Device: Investigational device

INTERVENTIONS:
Device: Investigational device — Device is an implantable neurostimulation system designed to deliver low-intensity electrical impulses to nerve structures.
  Other Names: St. Jude Medical Infinity™ Implantable Pulse Generator System (P140049), Deep Brain Stimulation (DBS) Directional Lead and Extension (P140009), Swift-Lock™ Anchor (K092371), Butterfly anchor (P140009)

SUMMARY:
Standard treatment options for patients who are diagnosed with BVFP include tracheostomy, cordotomy, arytenoidectomy, and suture tie-back. These standard treatment options may result in permanent damage to the vocal fold, therefore affecting the patient's ability to speak and compromising airway protection during swallowing. Additionally, these routine procedures cannot provide sufficient airway to permit significant aerobic activity. The goal in conducting this early feasibility study is to investigate the use of this device as a laryngeal pacemaker to treat BVFP.

DETAILED DESCRIPTION:
The recurrent laryngeal nerve (RLN) carries motor fibers that innervate both the abductor (PCA, opener) muscle and adductor (closer) muscles of the vocal folds. Damage to the nerve compromises both of these functions and arrests the vocal folds in a near-closed position. In case of BVFP, voice tends to be functional but airway embarrassment is often severe enough to warrant tracheostomy to relieve inspiratory stridor and dyspnea.

If spontaneous recovery from nerve injury does not occur within one year, it is likely the patient will be chronically paralyzed. In such instances, long-term tracheostomy could be considered. Unfortunately, permanent tracheostomy is known to have the complications of tracheal stenosis, chronic infection, and psycho-social impairment. For this reason, laryngeal surgery is offered to enlarge the airway and restore breathing through the mouth. These procedures, such as arytenoidectomy and cordotomy, where a portion of the larynx is surgically resected to enlarge the airway, also have inherent complications.

Although they represent the standard of care, they adversely affect voice and may compromise airway protection during swallowing. Further, they cannot provide sufficient airway to permit significant aerobic activity. The limitations associated with these current therapies have prompted investigation into a more physiologic, dynamic approach to rehabilitation: reanimation of the paralyzed PCA muscle by functional electrical stimulation (FES). Stimulation would be applied to the PCA muscle during the inspiratory phase of respiration to open the vocal folds. During noninspiratory phases, stimulation would cease and the vocal folds would passively relax to the midline to allow for normal voice production and airway protection in swallowing. Based on the research the investigators have conducted, the investigators expect patients would benefit from bilateral pacing through implantation of the neurostimulator by restoring normal ventilation, without negatively affecting the patient's voice or swallowing ability.

The investigators are collecting data in this study to show that this procedure is an effective means of a surgical approach for implantation of device with insertion and anchoring of the electrode leads. Incidence of complications both intraoperatively and postoperatively will also be collected and assessed. Any complications will be addressed according to current standard practice under the supervision of the operating surgeon. The device should produce an airway that will allow patients to breathe without a tracheostomy tube in place. Patients will be monitored for adverse events and managed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patients, 22 years of age or older
* Diagnosis of bilateral vocal fold paralysis, at least one year prior to study enrollment
* Must have tracheostomy in place minimum of 6 weeks prior to implantation of St.Jude Medical Infinity™ IPG device
* Demonstrated glottal opening bilaterally (abductory response) upon percutaneous needle stimulation of PCA muscles
* Demonstrated peak inspiratory flow with respiratory testing through the mouth of at least 0.4 L/sec

Exclusion Criteria:

* Any active illness that is associated with an immune disorder (such as diabetes)
* History of cardiac dysrhythmias or implanted cardiac pacemaker
* Any electronic implanted medical device that, in the investigator's opinion, could interact with the laryngeal pacemaker
* Active cardiac disease manifested by unstable angina, recent myocardial infarction, malignant arrhythmias, uncontrolled hypertension (diastolic greater than 110), or decompensated congestive heart failure
* Patients with underlying comorbidities that, in the investigator's opinion, could potentially warrant a need for oxygen therapy, including but not limited to: Chronic obstructive pulmonary disease, asthma, emphysema, recurrent bronchitis, pneumonia or interstitial lung disease
* Bilateral laryngeal immobility from stenosis or arthritis
* Poor Surgical risk patients as determined by the treating surgeon or Vanderbilt Preoperative Evaluation Center (VPEC)
* Patients with acute or chronic infections
* The abundance of interstitial fat may impede the surgical dissection. In the opinion of the principal investigator or treating physician(s), patients with factors that may complicate the surgical intervention will be excluded.
* Known allergy to barium dye or anesthetics
* Known allergy to any of the device materials
* Patients who in the opinion of the investigator, based on needle stimulation testing, have insufficient PCA muscle mass to implant leads
* Patients with pre-existing liquid dysphagia
* Presence of significant tracheal narrowing
* Any anatomical abnormality that would jeopardize safe implantation, per the treating surgeon
* Any medical condition, that in the opinion of the principal investigator or treating physician, would jeopardize the outcome or welfare of the participant
* Any history of keloid formation or hypertrophic scarring
* Females who are pregnant or plan a pregnancy within 1 year. A pregnancy test will be done as part of the routine pre-operative assessment for all females of childbearing potential.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Demonstration of a consistent surgical approach with successful implantation and functionality of a laryngeal pacemaker, as indicated by the presence of stimulated motion of the chronically paralyzed vocal fold. | 12 to 15 months

SECONDARY OUTCOMES:
Increased glottal area due to laryngeal pacemaker stimulation as assessed by increase in standard assessment testing. | 12 to 15 months
Increased ventilation due to laryngeal pacemaker stimulation as assessed by increase in standard assessment testing. | 12 to 15 months
Minimal impairment of voice due to laryngeal pacemaker stimulation as assessed by increase in standard assessment testing. | 12 to 15 months

CONTACTS AND LOCATIONS:
Overall Officials: David L. Zealear, PhD, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No